CLINICAL TRIAL: NCT03727074
Title: A Multi-Center, Double-Blind, Randomized, Vehicle-Controlled, Parallel-Group Bioequivalence Study to Compare Sol-Gel Technologies' 5-FU Cream, With Efudex® (5-FU) Cream, and Both Active Treatments to a Vehicle Control, in the Treatment of Actinic Keratosis
Brief Title: Bioequivalence Study to Compare Sol-Gel Technologies' 5-FU Cream With Efudex® (5-FU) Cream
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sol-Gel Technologies, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SGT-19-01
Record Dates: First submitted 2018-10-30; First posted 2018-11-01 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Actinic Keratosis (AK)
Keywords: Actinic Keratosis ,AK
MeSH Terms: conditions — Keratosis, Actinic | interventions — Fluorouracil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 5-FU Cream (Experimental): topical cream
  Interventions: Drug: 5-FU Cream
- Efudex® (Active Comparator): topical cream
  Interventions: Drug: Efudex®
- Vehicle (Placebo Comparator): topical cream
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: 5-FU Cream — topical cream twice a day
  Arms: 5-FU Cream
Drug: Efudex® — topical cream twice a day
  Arms: Efudex®
Drug: Vehicle — topical cream twice a day
  Arms: Vehicle

SUMMARY:
To compare the relative efficacy and safety and of 5-FU Cream to the marketed formulation Efudex® (5-FU) Cream, and to demonstrate the superior efficacy of the two active formulations over that of the Vehicle Control Cream, in the treatment of actinic keratosis.

DETAILED DESCRIPTION:
To compare the safety and efficacy profiles of 5-FU Cream with Efudex® (5-FU) Cream, and to demonstrate the superior efficacy of the two active formulations over that of the Vehicle Control Cream, in the treatment of actinic keratosis.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female 18 years of age and older.
2. Subject is able to understand and willing to sign Institutional Review Board (IRB) approved written informed consent for this study.
3. Subject must be generally healthy, based on medical records, and free from any clinically significant disease, other than AK, that in the opinion of the investigator might interfere with the study evaluations.
4. At least five (5) and no more than ten (10) clinically typical, visible or palpable, discrete AK lesions, each at least 4 mm in diameter on the face (excluding ears), forehead or bald scalp.

Exclusion Criteria:

1. Subject is pregnant, lactating, or is planning a pregnancy within the period of study participation.
2. Subject suffers from excessive alcohol consumption, drug abuse or has a condition that could compromise the subject's ability to comply with study requirements.
3. Presence of Atopic Dermatitis, Basal Cell Carcinoma, Eczema, Psoriasis, Rosacea, Squamous Cell Carcinoma or other possible confounding skin conditions on the

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
treatment success | week 6
  Proportion of subjects, in the Per-Protocol (PP) population, with treatment success, defined as complete clearing (100% clearance of all AK lesions within the designated treatment area) at the End of Study visit

CONTACTS AND LOCATIONS:
Locations (1):
- Core Healthcare Group, Cerritos, California, United States